CLINICAL TRIAL: NCT02341677
Title: SmartTarget - A Magnetic Resonance Image to Ultrasound Fusion System for Targeted Prostate Intervention: Biopsy
Brief Title: SmartTarget: BIOPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14/0044
Record Dates: First submitted 2014-11-24; First posted 2015-01-19 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Prostatic Neoplasms; Diagnostic Techniques and Procedures
Keywords: Prostatic Neoplasms; Diagnostic Techniques and Procedures; Magnetic Resonance Imaging; Ultrasonography; Biopsy; Image Fusion
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsy (Experimental): Single Arm Study. Biopsy Intervention.
  Interventions: Procedure: SmartTarget - Biopsy

INTERVENTIONS:
Procedure: SmartTarget - Biopsy — MRI to ultrasound fusion guided prostate biopsy

SUMMARY:
The purpose of this study is to determine how well SmartTarget guided prostate biopsies perform, compared with our current standard of "visually directed biopsies" in the detection of prostate cancer.

The diagnosis of prostate cancer is dependent upon sampling the prostate to confirm disease. Standard trans-rectal biopsies are taken in a random fashion, without prior knowledge of the disease location. Transperineal mapping biopsies overcome this by systematically samples the entire gland but are very intensive and time consuming to perform.

An alternative method is to perform targeted prostate biopsies where an MRI prior to biopsy can be used to inform doctors about the location of the disease. This is a difficult procedure to perform as it requires the surgeon to mentally translate the location of disease on MRI image to the live ultrasound seen in theatre.

SmartTarget may help this procedure by providing guidance to the location of the disease by fusing the MRI image onto the live ultrasound, thereby providing the clinician a target to biopsy.

This trial will compare the outcomes of "visually directed biopsies" with those directed by SmartTarget

ELIGIBILITY:
Inclusion Criteria:

* Previous TRUS biopsy with clinical indication for repeat biopsy
* Discrete lesion on mpMRI scoring 3, 4 or 5 on PI-RADs scale
* An understanding of the English language sufficient to understand written and verbal information about the trial and consent process
* Signed informed consent

Exclusion Criteria:

* Men who have taken any form of hormones (except 5-alpha reductase inhibitors) within the last 6 months
* Men with an irreversible coagulopathy predisposing to bleeding
* Men who are unability to undergo transrectal ultrasonography
* Men who have had previous radiation therapy to the pelvis
* Men who have had HIFU, cryosurgery, thermal, irreversible electroporation, photodynamic, photothermal therapy, or microwave therapy to the prostate. Transurethral resection or vaporization of the prostate for benign prostatic hyperplasia using any energy modality is permitted
* Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
* Men who are unable to give informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cancer Detection | Within 3 weeks of biopsy
  The proportion of men with clinically significant disease based on SmartTarget guided biopsy compared to the proportion of men with clinically significant disease based on visually-directed biopsy.

SECONDARY OUTCOMES:
Targeting Efficiency (core length, grade) | Within 3 weeks of Biopsy
  The targeting efficiency of the SmartTarget guided biopsies versus visually-directed biopsies measured by:
  Number of cores required to obtain the highest cancer risk category Number of cores with cancer Maximum Cancer Core Length and Total Cancer Core Length Highest Grade Cancer
Clinical Usability (length of procedure, generation time, re-registration rate, failure rate) | During Procedure
  To evaluate the clinical usability of SmartTarget guided biopsy as measured by:
  Length of Procedure SmartTarget model generation time SmartTarget re-registration rate SmartTarget failure rate
Quality of Life | 6 Weeks post biopsy
  To assess how this biopsy strategy impacts on quality of life as measured using validated questionnaires:
  IPSS IIEF EQ5D - 5L

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, FRCS PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom